CLINICAL TRIAL: NCT00986440
Title: A Randomized, Double-Blind Placebo-Controlled Phase 2 Study of CS-7017 in Colorectal Cancer Patients Who Have Achieved Disease Control Following First-Line Chemotherapy
Brief Title: Study of CS-7017 in Colorectal Cancer Patients Who Have Achieved Disease Control Following First-Line Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to changes to the standard of care within the proposed market for CS-7017.
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CS7017-A-E201
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Results first posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — efatutazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CS-7017 (Experimental)
  Interventions: Drug: CS-7017
- Placebo (Placebo Comparator): Placebo matching CS-7017
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CS-7017 — CS-7017
  Arms: CS-7017
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Monotherapy treatment with CS-7017 to assess progression-free-survival (PFS) of subjects who achieved an objective response of Disease Control on first line therapy with Folinic acid (leucovorin), Fluorouracil (5-FU), Oxaliplatin (Eloxatin) known as FOLFOX; or Folinic acid (leucovorin), Fluorouracil (5-FU), irinotecan (Camptosar) known as FOLFIRI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed, metastatic CRC that have achieved confirmed maximal benefit of DC following treatment with standard first line chemotherapy of a 5-fluoropyrimidine plus either oxaliplatin or irinotecan. Patients should be entered onto this trial within 8 weeks of completing first line therapy;
* If CR was not achieved: measurable disease, i.e. at minimum one unidimensionally-measurable target lesion according to RECIST (Response Evaluation Criteria in Solid Tumors);
* Age >= 18 years and Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 2 at study entry;
* Resolution of any toxic effects of prior therapy (except alopecia) to NCI CTCAE, Version 3.0, grade =< 1;
* Adequate organ and bone marrow function as evidenced by:

  * Haemoglobin >= 10 g/dL (transfusion and/or growth factor support allowed);
  * Absolute neutrophil count (ANC) >= 1.5 x 109/L;
  * Platelet count >= 100 x 109/L;
  * Serum creatinine =< 1.5 x ULN or creatinine clearance >60 mL/min;
  * AST and alkaline phosphatase <2.5 x ULN if without liver metastasis and =< 5.0 x ULN if liver metastasis;
  * Total bilirubin =< 2.0 x ULN;
  * Prothrombin time (PT)/International Normalised Ratio (INR) within normal limits (WNL) unless therapeutically anticoagulated;
* Women of childbearing potential and men must be willing to consent to using highly effective methods of contraception (eg, hormonal contraceptives, bilateral tubal ligation, barrier with spermicide, intrauterine device) while on treatment and for at least 3 months thereafter;
* Males with the potential to father children must use two of the following methods of contraception acceptable for the study (e.g. hormonal contraceptives, bilateral tubal ligation, barrier with spermicide, intrauterine device) while on trial treatment and for at least 3 months thereafter.
* All female subjects of childbearing potential must have a negative pregnancy test (plasma or urine) result within 7 days before initiating study treatment;
* Baseline laboratory tests and tumor assessments must have been performed within 2 weeks before initiating study treatment;
* Subjects must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects) and must sign and date an IEC-approved ICF before performance of any study specific procedures or tests.

Exclusion Criteria:

* Anticipation of need for a major surgical procedure or RT during the study;
* Treatment with chemotherapy, hormonal therapy, minor surgery, or any investigational agent within 4 weeks before study enrolment. Treatment with immunotherapy, biological therapy, or major surgery within 6 weeks before study enrolment. Treatment with RT within 1 week before study enrolment.
* History of any of the following conditions: diabetes mellitus requiring treatment with insulin or oral agents;
* Concomitant use of other TZDs;
* Myocardial infarction with significant impairment of cardiac function (e.g., ejection fraction =< 50%); severe/unstable angina pectoris; coronary/peripheral artery bypass graft; congestive heart failure; cerebrovascular accident (CVA) or transient ischemic attack (TIA), pulmonary embolism, or other clinically significant thromboembolic event; clinically significant pulmonary disease (e.g., severe chronic obstructive pulmonary disease [COPD] or asthma);
* Brain metastasis; an uncontrolled seizure disorder; spinal cord compression; or carcinomatous meningitis;
* Pleural or pericardial effusion. Subjects with minimal pleural effusion may be eligible upon request by Investigator and approval by Sponsor;
* Clinically significant active infection that requires antibiotic therapy or Human Immunodeficiency Virus (HIV) positive subjects receiving antiretroviral therapy;
* Pregnant or breast feeding;
* Known history of severe hypersensitivity reactions to any of the components of CS 7017 formulations;
* Serious intercurrent medical or psychiatric illnesses or any other conditions that in the opinion of the Investigator would impair the ability to give informed consent or unacceptably reduce protocol compliance or safety of the study treatment;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-07-31 (Actual); Primary Completion 2012-10-29 (Actual); Study Completion 2012-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (39):
- Czechia (3):
  - Fakulti nemocnice Brno, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Nemocnice Znojmo, p.o., Oddeleni radiacni a klinicke onkologie, Znojmo
- France (4):
  - Hopitaux civils de colmar, Colmar, Cedex
  - Hopital Edouard Herriot, Lyon, Cedex
  - Service d'Oncologie Medicale, Rennes, Cedex
  - Centre Hospitalier Prive Saint Gregoire, Saint-Grégoire
- Germany (3):
  - Onkologische Praxis Donauwörth, Donauwörth
  - Universitätsklinikum Halle Klinik und Poliklinik für Innere Medizin, Halle
  - Klinikum rechts der Isar, München
- Italy (5):
  - Institute for Cancer Research and Treatment - IRCC, Candiolo, Torino
  - Ospedale San Martino, Genova
  - Unita Operativa di Oncologia Medica, Lecce
  - Policlinico Santa Maria alle Scotte, Siena
  - Azienda Ospedaliero Universitaria Santa Maria della Misericordia, Udine
- Poland (5):
  - Bialostockie Centrum Onkologii im. Marii Sklodowskiej-Curie w Bialymstoku, Bialystok
  - Wojewodzki Szpital Specjalistyczny, Bytom
  - Centrum Onkologii Instytut im. Marii Sklodowskiej-Curie, Gliwice
  - VESALIUS Sp. z o.o., Krakow
  - NZOZ ONKOLOG s.c., Warsaw
- Russia (8):
  - Medical Radiological Research Centre, Obninsk, Kaluga Oblast
  - Kazan State Medical University, Kazan', Tatarstan Republic
  - Russian Oncology Research Centre n.a. Blokhin, RAMS, Moscow
  - Central Clinical Hospital #1, Moscow
  - NUZ Semashko Central Clinical Hospital, Moscow
  - Federal State Institution of Healthcare Clinical Hospital # 122 n.a.L.G Sokolov, Saint Petersburg
  - St-Petersburg State Institution of Public Health, Saint Petersburg
  - Tula Regional Oncology dispensary, Tula
- Spain (3):
  - H.Clinic I Provincial de Barcelona, Barcelona, Villaroel
  - Clinica Universitaria de Navarra, Pamplona
  - Hospital Mútua de Terrassa, Terrassa (Barcelona)
- Ukraine (3):
  - Volyn regional oncology dispensary, Lutsk, Volyn Oblast
  - Kyiv City Oncology Hospital, Kiev
  - Sumy Regional Oncology Center, Sumy
- United Kingdom (5):
  - Mount Vernon Cancer Centre, Northwood, Middlesex
  - Aberdeen Royal Infirmary, Aberdeen
  - St.Bartholomew's Hospital, London
  - UCLH Cancer Clinical Trials Unit, London
  - Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 84 participants who met all inclusion criteria and no exclusion criteria were enrolled at 46 clinic sites in Europe. Of the 84 participants enrolled, 83 received treatment.
Pre-assignment Details: Participants who were randomized to treatment (CS-7017 0.5 mg or placebo) started treatment within 8 weeks of completing first-line therapy.
Groups:
- CS-7017 0.5 mg: Participants who were randomized to receive two 0.25 mg CS-7017 tablets (i.e. a dose of 0.5 mg) administered by mouth twice daily (PO BID), for a total of four tablets per day.
- Placebo: Participants who were randomized to receive matching placebo.
Period: Overall Study
Arm/Group | CS-7017 0.5 mg | Placebo
Started | 41 | 43
Randomized, But Not Dosed | 0 | 1
Completed | 0 | 0
Not Completed | 41 | 43
Not completed — Progressive disease | 27 | 37
Not completed — Serious adverse event or adverse event | 9 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Screen failure (not dosed) | 4 | 2

BASELINE CHARACTERISTICS:
Population: The demographics and baseline characteristics were based on the intent-to-treat analysis set.
Groups:
- Total: Total of all reporting groups
Arm/Group | CS-7017 0.5 mg | Placebo | Total
Number analyzed (Participants) | 41 | 43 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (7.69) | 60.9 (9.73) | 62.4 (8.88)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 24 | 26 | 50
  ≥65 years | 17 | 17 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 22 | 24 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 40 | 41 | 81
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage Rate of Progression-free Survival at 18 Weeks Following Use of CS-7017 in Colorectal Cancer Participants Who Have Achieved Disease Control Following First-Line Chemotherapy
Description: Progression-free survival (PFS) was defined as the time from enrollment to the date of the first objective documentation of disease progression or death resulting from any cause, whichever comes first. Progression was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) as at least a 20% increase in the sum of diameters of target lesions.
Time Frame: 18 weeks postdose
Population: PFS was assessed in the Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CS-7017 0.5 mg | Placebo
Number analyzed (Participants) | 39 | 42
percentage of participants | 39.86 [23.5 to 55.7] | 25.00 [13.0 to 39.0]
Statistical Analysis 1: Comparison: CS-7017 0.5 mg vs Placebo; Test type: Superiority; p < 0.0001, 2-sided P value for z test; Z statistic for difference = 3.92
Statistical Analysis 2: Comparison: CS-7017 0.5 mg vs Placebo; Test type: Superiority; Hazard Ratio, log = -0.41

2. Secondary Outcome: Percentage Rate of Progression-free Survival Following Use of CS-7017 in Colorectal Cancer Participants Who Have Achieved Disease Control Following First-Line Chemotherapy
Description: as for outcome 1
Time Frame: At 12, 24, and 30 weeks postdose
Population: PFS was assessed in the Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CS-7017 0.5 mg | Placebo
Number analyzed (Participants) | 39 | 42
percentage of participants
  Progression-free survival at 12 weeks | 62.0 [44.6 to 75.5] | 47.5 [31.6 to 61.8]
  Progression-free survival at 24 weeks | 29.9 [15.4 to 45.9] | 15.0 [6.1 to 27.6]
  Progression-free survival at 30 weeks | 29.9 [15.4 to 45.9] | 12.5 [4.6 to 24.6]
Statistical Analysis 1: Comparison: CS-7017 0.5 mg vs Placebo; Test type: Superiority; p = 0.0380, Log Rank
Statistical Analysis 2: Comparison: CS-7017 0.5 mg vs Placebo; Test type: Superiority; p = 0.1773, Peto-Peto-Prentice
Statistical Analysis 3: Comparison: CS-7017 0.5 mg vs Placebo; Test type: Superiority; p = 0.2844, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: CS-7017 0.5 mg vs Placebo; Test type: Superiority; p = 0.1140, Tarone-Ware

3. Secondary Outcome: Percentage Rate of Overall Survival Following Use of CS-7017 in Colorectal Cancer Participants Who Have Achieved Disease Control Following First-Line Chemotherapy
Description: Overall survival (OS) was defined as the time from the date of enrollment to the date of death and assessed by Kaplan Meier analysis.
Time Frame: At 3, 6, 9, and 12 months postdose
Population: OS was assessed in the Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CS-7017 0.5 mg | Placebo
Number analyzed (Participants) | 39 | 42
percentage of participants
  Overall survival rate at 3 months | 100.0 [100.0 to 100.0] | 92.9 [79.5 to 97.6]
  Overall survival rate at 6 months | 87.2 [71.9 to 94.5] | 85.5 [70.4 to 93.2]
  Overall survival rate at 9 months | 74.4 [57.6 to 85.3] | 75.2 [58.7 to 85.8]
  Overall survival rate at 12 months | 68.4 [51.0 to 80.7] | 55.4 [37.2 to 70.3]
Statistical Analysis 1: Comparison: CS-7017 0.5 mg vs Placebo; Test type: Superiority; p = 0.1213, Log Rank

4. Secondary Outcome: Best Overall Response and Objective Response Rate Following Use of CS-7017 in Colorectal Cancer Participants Who Have Achieved Disease Control Following First-Line Chemotherapy
Description: The best overall response was defined as the best response (in the order of confirmed complete response [CR], confirmed partial response [PR], unconfirmed CR, unconfirmed PR, stable disease [SD], and progressive disease [PD]) among all overall responses recorded from the start of treatment until the participant withdrew from the study. If there was no tumor assessment after the first dose of study drug, the best overall response was classified as Inevaluable. Based on RECIST v1.0, CR was defined as a disappearance of all target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target lesions, and SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target lesions.
Time Frame: From baseline up to disease progression or the development of unacceptable toxicity (whichever occurs first), up to approximately 3 years 3 months
Population: Best overall response and objective response rate were assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | CS-7017 0.5 mg | Placebo
Number analyzed (Participants) | 39 | 42
Participants
  Confirmed CR | 5 | 1
  Confirmed PR | 1 | 0
  Objective response (confirmed CR+PR) | 6 | 1
  Unconfirmed CR | 0 | 0
  Unconfirmed PR | 0 | 3
  Stable disease | 10 | 8
  Progressive disease | 20 | 27
  Inevaluable | 3 | 3
  Best overall response of SD or better | 16 | 12

5. Secondary Outcome: Duration of Response for Responding Participants Following Use of CS-7017 in Colorectal Cancer Participants Who Have Achieved Disease Control Following First-Line Chemotherapy
Description: Duration of response was defined for participants with confirmed CR or PR and confirmed and unconfirmed CR or PR as the time from the date of the first documentation of objective response (CR or PR) to the date of the first documentation of progressive disease. Duration of SD was defined for participants whose best response was SD as the time from the randomization date to the date of the first documentation of progressive disease. Duration of response was estimated using Kaplan Meier methods.
Time Frame: From the date of first objective response (confirmed and unconfirmed CR or PR) to date of progressive disease, up to 3 years 3 months
Population: Duration of response was assessed in the Full Analysis Set. Number Analyzed for each Row represents only the participants with CR or PR (confirmed and unconfirmed) and SD.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | CS-7017 0.5 mg | Placebo
Number analyzed (Participants) | 39 | 42
weeks
  Duration of response (confirmed responses): number analyzed (Participants) | 6 | 1
  Duration of response (confirmed responses) | 33.57 (25.88) | 37.86 (NA) — SD could not be calculated on a single participant.
  Duration of response (confirmed and unconfirmed): number analyzed (Participants) | 6 | 4
  Duration of response (confirmed and unconfirmed) | 33.57 (25.88) | 15.96 (14.86)
  Duration of stable disease: number analyzed (Participants) | 10 | 8
  Duration of stable disease | 26.16 (10.68) | 22.52 (8.01)

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events Related to Study Drug With an Incidence of ≥5% Following Use of CS-7017 Or Placebo in Colorectal Cancer Participants Who Have Achieved Disease Control Following First-Line Chemotherapy
Description: A treatment-emergent adverse event (TEAE) was defined as any untoward, unfavorable, unintended medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event that occurs more than 30 days after the last dose of study medication is not included as a TEAE unless it is considered related to treatment. If relationship is missing, the AE is also considered to be related to the drug.
Time Frame: Baseline up to 30 days after last study dose, up to 3 years 3 months
Population: Adverse events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | CS-7017 0.5 mg | Placebo
Number analyzed (Participants) | 41 | 42
Participants
  Any Related TEAE | 37 | 16
  Any Blood and Lymphatic System Disorder | 7 | 0
  Anaemia | 6 | 0
  Any General Disorder& Administration Site Disorder | 23 | 6
  Face oedema | 4 | 1
  Fatigue | 6 | 3
  Localised oedema | 3 | 0
  Oedema | 3 | 0
  Oedema peripheral | 16 | 2
  Any Gastrointestinal Disorder | 6 | 2
  Any Investigations | 22 | 7
  Weight increased | 20 | 5
  Any Metabolism and Nutrition Disorder | 6 | 3
  Fluid retention | 5 | 2
  Any Respiratory, Thoracic, & Mediastinal Disorder | 8 | 0
  Dyspnoea | 4 | 0
  Pleural effusion | 3 | 0
  Any Skin and Subcutaneous Tissue Disorder | 5 | 3

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from baseline up to 30 days after last dose, up to 3 years 3 months in the Safety Analysis Set.
Description: A TEAE was defined as any untoward, unfavorable, unintended medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An adverse event that occurs more than 30 days after the last dose of study medication is not included as a TEAE unless it is considered related to treatment. If relationship is missing, the AE is also considered to be related to the drug.
Arm/Group | CS-7017 0.5 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 16/41 | 23/42
Serious Adverse Events (participants affected / at risk) | 6/41 | 5/42
Other Adverse Events (participants affected / at risk) | 41/41 | 31/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CS-7017 0.5 mg (N=41) | Placebo (N=42)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CS-7017 0.5 mg (N=41) | Placebo (N=42)
Anaemia (Blood and lymphatic system disorders) | 15 | 0
Tachycardia (Cardiac disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 9
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 7
Nausea (Gastrointestinal disorders) | 5 | 5
Proctalgia (Gastrointestinal disorders) | 0 | 4
Asthenia (General disorders) | 10 | 2
Face oedema (General disorders) | 4 | 1
Fatigue (General disorders) | 11 | 6
Localised oedema (General disorders) | 3 | 0
Oedema (General disorders) | 3 | 1
Oedema peripheral (General disorders) | 17 | 2
Pyrexia (General disorders) | 2 | 3
Weight increased (Investigations) | 21 | 5
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3
Fluid retention (Metabolism and nutrition disorders) | 5 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4
Dizziness (Nervous system disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
Early termination was due to changes in the standard of care within the proposed market. The study was designed when patient monitoring and no treatment was an option that will not support a confirmatory Phase 3 study. No safety or efficacy concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No